CLINICAL TRIAL: NCT00808262
Title: A Phase I/II, Open-label, Escalating Dose, "Optimal Two-stage", Study of TNFα-Kinoid (TNF- K) Immunization in Crohn's Disease Patients
Brief Title: Safety and Immunogenicity of a TNFa Kinoid in Patients With Crohn's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Neovacs (Industry)
Responsible Party: Pierre Vandepapeliere, CMO, Neovacs SA
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TNF-K-001
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Crohn's Disease
Keywords: anti-TNFa; immunization; kinoid; crohn's disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TNFa Kinoid dose 1 (Experimental)
  Interventions: Biological: TNFa Kinoid
- TNFa Kinoid dose 2 (Experimental)
  Interventions: Biological: TNFa Kinoid
- TNFa Kinoid dose 3 (Experimental)
  Interventions: Biological: TNFa Kinoid

INTERVENTIONS:
Biological: TNFa Kinoid — TNFa kinoid at days 0, 7, 28

SUMMARY:
Evaluation of the safety and the immune response induced by active immunization through a TNFa kinoid in patients with Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have Active Crohn's Disease, as defined by a Crohn's Disease Activity Index (CDAI) score of >220 but ≤400, with active Crohn's disease of ileum and/or colon (Other areas may be involved if ileum and/or colon are also involved)based upon either endoscopic, histologic and/or radiographic evidence
* Patients with active disease despite treatment with 5-ASAs or sulfasalazine, corticosteroids (prednisone, budesonide, other), AZA or 6-MP or cyclosporine or MTX or Tacrolimus, ; OR intolerant of 5-ASAs or sulfasalazine; or intolerant of antibiotics; or intolerant of corticosteroids (prednisone, budesonide, other); or intolerant of AZA or 6-MP or cyclosporine or MTX or Tacrolimus
* Patients might have previously responded to any prior anti-TNF agents and then lost response OR might be intolerant of any prior anti-TNF agents
* Positive skin reaction to challenge with Candida antigens
* Written informed consent

Exclusion Criteria:

* Prior history of tuberculosis or positive chest X ray or positive purified protein derivative skin test or positive interferon gamma TB assay
* Signs or symptoms of clinically significant stricture of bowel.
* Total parenteral nutrition or elemental diet required for treatment of disease or support of short bowel syndrome
* Presence of an enteric stoma
* Imminent or urgent surgery required for infection, abscess, bleeding or any other cause relating to their Crohn's Disease or other condition
* History of malignancy. However, subjects with basal call carcinomas or less than 3 squamous cell carcinomas are allowed
* History of asthma or serious allergic condition (including history of seafood allergy)
* Serious local infection (e.g., cellulitis, abscess) or systemic infection (e.g., pneumonia, septicemia) within the 3 months prior to the first dose of study drug
* History of opportunistic infection excluding oral candidiasis on steroids
* Enteric infection as evidenced by positive stool C&S, O&P and C. difficile obtained during screening
* Any significant or decompensated cardiac, neurologic, liver, pulmonary or renal disease
* History of lymphoproliferative disorders
* Clinically significant abnormal hematology values, as determined by the investigator, for hematocrit, hemoglobin, white blood cell count or platelets
* Clinically significant abnormal blood chemistry values as determined by the investigator
* Current significant drug or alcohol abuse as determined by the investigator
* Positive for hepatitis C antibody or positive for hepatitis B surface antigen (HbsAg) or HIV infection
* Surgery within the previous 3 months (other than minor cosmetic surgery or minor dental procedures)
* Participation in a clinical study (including previous participation in this study) within the previous 4 months
* Had a primary non-response to any prior anti-TNF agents as defined by the investigator OR received any prior anti-TNF agents within the past 8 weeks prior to study entry
* Pregnancy and lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | Whole study period

SECONDARY OUTCOMES:
Antibody response | Day 38

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Vandepapeliere, MD, PhD, Study Director — Neovacs
Locations (6):
- South Africa (4):
  - Durbanville Medi-Clinic, Cape Town, Cape
  - Parexel Port Elizabeth, Port Elizabeth, Eastern Cape
  - Farmovs Parexel, Bloemfontein
  - Parexel George, George
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Universitätsspital Zürich, Zurich